CLINICAL TRIAL: NCT05559918
Title: Dual-antiplatelet Therapy Strategies for Elective PCI in a Real-world Setting
Acronym: DAPT-FOR-REAL
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Ronak Delewi, Principal Investigator Dr. R Delewi, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: AUMC25485
Record Dates: First submitted 2022-09-21; First posted 2022-09-29 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
Keywords: Pretreatment; Diagnostic angiography; ad-hoc PCI
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Preloading with clopidogrel
- In-hospital loading with clopidogrel

SUMMARY:
To assess the safety and efficacy of in-laboratory clopidogrel loading dose administration before ad-hoc PCI versus clopidogrel preloading treatment in patients planned for diagnostic angiography with optional ad-hoc PCI.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women aged at least 18 years
* Scheduled for diagnostic CAG due to suspected obstructive coronary artery disease

Exclusion Criteria:

* Presence of contra-indications for the use of clopidogrel (hypersensitivity or known allergy to clopidogrel, severe liver insufficiency, resent or active pathological bleeding, patients known to be poor CYP2C19 metabolizers, patients using pharmacological CYP2C19 inhibitors and inducers)
* Patients using clopidogrel for other reasons than the scheduled diagnostic CAG (e.g. due to previous stroke)
* Patients using P2Y12 inhibitors other than clopidogrel (e.g. prasugrel, ticagrelor, cangrelor)
* Patients using VKA (e.g. acenocoumarol, fenprocoumon)
* Patients using DOAC/NOAC (e.g. apixaban, dabigatran, edoxaban, rivaroxaban)
* Inability to give informed consent (e.g., language barrier)
* Patients who have a documented mentioning of previous denial to any trial participation in the electronic patient dossier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients aged 18 years and older who have been referred for diagnostic CAG due to symptoms suggestive of obstructive coronary artery disease with optional ad-hoc PCI.
Sampling Method: Probability Sample
Enrollment: 1462 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Net adverse clinical events (NACE) | 30 days
  The incidence rate of NACE (the composite of the clinical events all-cause death, myocardial infarction, definite/probable stent thrombosis, stroke and BARC type 2, -3 or -5 bleeding) wil be compared between groups at 30 days

SECONDARY OUTCOMES:
Bleeding (classified as BARC type 2, -3 and -5 bleeding) | In-hospital, at 30 days
  The incidence rate of bleeding (classified as BARC type 2, -3 and -5 bleeding) will be compared between groups
Patient oriented clinical events (POCE) | In-hospital, at 30 days
  The incidence rate of POCE (the composite of clinical events all-cause death, stroke, myocardial infarction, and repeat revascularization) will be compared between groups
All-cause mortality | In-hospital, at 30 days
  The incidence rate of all-cause mortality will be compared between groups
Myocardial infarction | In-hospital, at 30 days
  The incidence rate of myocardial infarction will be compared between groups
Stent thrombosis (definite/probable) | In-hospital, at 30 days
  The incidence rate of stent thrombosis (definite and probable) will be compared between groups
Stroke | In-hospital, at 30 days
  The incidence rate of stroke will be compared between groups
Repeat revascularisation | In-hospital, at 30 days
  The incidence rate of repeat revascularisation will be compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Ronak Delewi, MD, PhD, Principal Investigator — Amsterdam University Medical Center, location AMC
Locations (2):
- Netherlands (2):
  - Amsterdam Universitair Medisch Centrum (AUMC) - Locatie AMC, Amsterdam, North Holland
  - Amsterdam Universitair Medisch Centrum (AUMC) - Locatie VUMC, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: No